CLINICAL TRIAL: NCT04324645
Title: Active Symptom Monitoring in Patients Undergoing Radiation Therapy for Thoracic Malignancies
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Other Study IDs: 202003007
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Symptom Monitoring; Radiation Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active Symptom Monitoring via Noona: Participants will undergo a single training session on how to use the Noona software no more than 4-12 weeks before starting therapy. They can start using the software immediately after the training session. Patients will be invited to complete either the Chest Radiotherapy (if radiotherapy alone), Chemotherapy-18 (if chemoradiation therapy), or Bone Radiotherapy (if other) module at baseline, every other week throughout therapy, and during follow up for 90-days. Patients will be encouraged by the treatment team to complete the baseline symptom report prior to starting any therapy and to complete the reports during therapy and in follow up. Patients will also complete the EORTC QLQ-C30 and the NCCN Distress Thermometer at baseline (no more than 12 weeks before starting therapy), within 1 week of completing therapy, and at 90-days follow up. Patients will be encouraged to use Noona's other features beyond invited modules and PRO inventories, such as the diary during the study
  Interventions: Other: Noona Software

INTERVENTIONS:
Other: Noona Software — Enrolled patients will be provided with login information for their Noona account. Patients will log in to the Noona symptom monitoring system using their own computer hardware. Any type of personal computer or compatible mobile device will be allowed (i.e. iPhone, Android phone). Patients will be able to access the Noona system from any internet access point and will be provided with the hospital/clinic public WiFi information.

SUMMARY:
This study seeks to achieve two aims:

* To assess the implementation of Noona software for continuous symptom monitoring for a diverse population of patients with thoracic malignancies who are undergoing radiation and
* To validate remote collection of standardized PRO measures using Noona software.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed cancer. Radiographically apparent (i.e. not histologically or cytologically confirmed) malignancy of the thorax is allowed.
* Currently planning to receive radiotherapy with or without chemotherapy for greater than one fraction.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).
* Age 18 years or older

Exclusion Criteria:

-Unable to reliably access and use a device compatible with Noona software.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a single-site study, which will be open at Siteman Cancer Center at Washington University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2022-03-13 (Actual); Study Completion 2022-03-13 (Actual)

PRIMARY OUTCOMES:
Percentage of invited symptom reports completed during the study period | Treatment through 90 days of follow-up (estimated to be 5 months)
Percentage of questions completed within each invited symptom report | Treatment through 90 days of follow-up (estimated to be 5 months)

SECONDARY OUTCOMES:
Patient reported outcomes as measured by EORTC QLQ-C30 | Baseline, within 1 week of completing therapy and at 90-day follow-up
  It includes five function domains (physical, emotional, social, role, cognitive), eight symptoms (fatigue, pain, nausea/vomiting, constipation, diarrhea, insomnia, dyspnea, and appetite loss), as well as global health/quality-of-life and financial impact. Patients respond on a four-point scale from "not at all" to "very much" for most items. Most items use a "past week" recall period. Raw scores are linearly converted to a 0-100 scale with higher scores reflecting higher levels of function and higher levels of symptom burden.
Patient reported outcomes as measured by NCCN Distress Thermometer | Baseline, within 1 week of completing therapy and at 90-day follow-up
  Measures distress experienced during the past week. 10 = extreme distress and 0=no distress

CONTACTS AND LOCATIONS:
Overall Officials: Matthew B Spraker, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu